CLINICAL TRIAL: NCT04523571
Title: Safety and Immunogenicity of SARS-CoV-2 mRNA Vaccine (BNT162b1) in Chinese Healthy Subjects: A Phase I, Randomized, Placebo-controlled, Observer-blind Study
Brief Title: Safety and Immunogenicity of SARS-CoV-2 mRNA Vaccine (BNT162b1) in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BNT162-03
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: SARS-CoV-2
Keywords: Protection against COVID-19; Coronavirus Disease 2019; Coronavirus infection; Vaccine; RNA Vaccine; Virus Diseases
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Virus Diseases | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Low-dose, 18-55 years of age (Experimental)
  Interventions: Biological: BNT162b1
- High-dose, 18-55 years of age (Experimental)
  Interventions: Biological: BNT162b1
- Placebo, 18-55 years of age (Placebo Comparator)
  Interventions: Other: Placebo
- Low-dose, 65-85 years of age (Experimental)
  Interventions: Biological: BNT162b1
- High-dose, 65-85 years of age (Experimental)
  Interventions: Biological: BNT162b1
- Placebo, 65-85 years of age (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BNT162b1 — Intramuscular injection
  Arms: High-dose, 18-55 years of age; High-dose, 65-85 years of age; Low-dose, 18-55 years of age; Low-dose, 65-85 years of age
Other: Placebo — Intramuscular injection
  Arms: Placebo, 18-55 years of age; Placebo, 65-85 years of age

SUMMARY:
This was a phase I, randomized, placebo-controlled, observer-blind study, for evaluation of safety and immunogenicity of SARS-CoV-2 mRNA vaccine (BNT162b1) in Chinese healthy population.

DETAILED DESCRIPTION:
The participants were screened for 2 weeks (Day -14 to Day 0) before randomization, and received 1 dose of SARS-CoV-2 vaccine (BNT162b1) or placebo intramuscularly (IM) on Day 1 and Day 22, respectively. After randomization, the study for each participant lasted for approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

For adult group (age ≥18 and ≤55)

* Male or female subjects of ≥18 years old and ≤55 years old with body mass index (BMI) ≥18 and ≤30 at the Screening Visit.
* Individuals who are in good health condition at the time of entry into the trial as determined by medical history, physical examination (including vital signs, electrocardiogram [ECG]) and eligibility screening test (hematology, blood chemistry and urine analysis) and clinical judgment of the investigator at Screening Visit.
* The subject can provide with informed consent and signs and dates a written informed consent form (ICF) prior to the initiation of any trial procedures.
* They must be able to understand and follow trial-related instructions.
* They must be willing and able to comply with planned visits, treatment schedule, laboratory tests and other requirements of the trial.
* Negative in antibodies screening of SARS-CoV-2 (fingerstick).
* Normal in chest computed tomography (CT) scans (no imaging features of COVID-19).
* Axillary temperature ≤ 37.0ºC.
* Negative SARS-CoV-2 test in throat swabs by reverse transcription-polymerase chain reaction (RT-PCR).
* Women of childbearing potential (WOCBP) must have a negative beta-human chorionic gonadotropin (β-hCG) in serum sample at Screening Visit. Women that are postmenopausal (Menopause≥12 consecutive months) or permanently sterilized will be considered as not having reproductive potential.
* WOCBP must have used effective contraception 14 days prior to screening and agree to use effective contraception continuously during the trial period, from 14 days prior to Screening Visit to 60 days after the last immunization.
* WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during trial, starting from Screening Visit and continuously until 60 days after being given the last immunization.
* Men who are sexually active with a WOCBP and have not had a vasectomy must agree to practice an effective form of contraception with their female partner of childbearing potential during the trial, starting from Screening Visit and continuously until 60 days after being given the last immunization.
* Men must be willing to refrain from sperm donation, starting from Screening Visit and continuously until 60 days after receiving the last immunization.

For the elderly group (age ≥65 and ≤85)

* Male or female subjects ≥65 years old and ≤85 years old at Screening Visit
* Individuals who are in a health condition that can receive the investigational vaccine, at the time of entry into the trial as determined by medical history, physical examination (including vital signs, ECG) and eligibility screening tests (hematology, biochemistry and urinalysis) and clinical judgment of the investigator at Screening Visit.
* The subject can provide with informed consent and signs and dates a written ICF prior to the initiation of any trial procedures.
* They must be able to understand and follow trial-related instructions.
* They must be willing and able to comply with planned visits, treatment schedule, laboratory tests and other requirements of the trial.
* Negative in antibodies screening of SARS-CoV-2 (blood sample from fingertip).
* No imaging features of COVID-19 in chest CT.
* Axillary temperature ≤ 37.0ºC.
* Negative SARS-CoV-2 test in throat swabs by RT-PCR.
* WOCBP must have a negative serum β-hCG at Screening Visit. Women that are postmenopausal (Menopause ≥12 consecutive months) or permanently sterilized will be considered as not having reproductive potential.
* WOCBP must have used effective contraception 14 days prior to screening and agree to use effective contraception continuously during the trial period, from 14 days prior to Screening Visit to 60 days after the last immunization.
* WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during trial, starting from Screening Visit and continuously until 60 days after being given the last immunization.
* Men who are sexually active with a WOCBP and have not had a vasectomy must agree to practice an effective form of contraception with their female partner of childbearing potential during the trial, starting from Screening Visit and continuously until 60 days after being given the last immunization.
* Men must be willing to refrain from sperm donation, starting from Screening Visit and continuously until 60 days after receiving the last immunization.

Exclusion Criteria:

For adult group (age ≥18 and ≤55)

* Have had any acute illness, as determined by the investigator, with or without fever, within 72 hours prior to the prime vaccination. An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the investigator, the residual symptoms will not compromise their well-being if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
* Are breastfeeding on the day of Screening Visit or who plan to breastfeed during the trial, starting from Screening Visit and continuously until at least 90 days after the last immunization. Women or partners who plan to become pregnant within 1 year post the Screening Visit.
* Have a known allergy, hypersensitivity, or intolerance to the planned vaccine for trial including any excipients.
* Used to have a history of hypersensitivity or serious reactions to vaccination.
* Received any vaccination within 4 weeks prior to Visit 1.
* Don't agree to not be vaccinated during the trial, starting from Screening Visit and continuously until 28 days after receiving the last immunization, except emergency vaccination (e.g. rabies vaccine, tetanus vaccine).
* Had any medical condition (e.g., autoimmune disease) or any major surgery (e.g., requiring general anesthesia) within the past 5 years, which in the opinion of the investigator, could compromise their well-being if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
* Have any surgery planned during the trial, starting from Screening Visit and continuously until at least 90 days after the last immunization.
* Had any chronic use (more than 14 continuous days) of any systemic medications that affects immune function, including immunosuppressant or other immune-modifying drugs, within 6 months prior to Screening Visit unless in the opinion of the investigator, the medication would not prevent, limit, or confound the protocol-specified assessments or could compromise safety of subjects.
* Had administration of any immunoglobulins and/or any blood products within the 3 months prior to Screening Visit.
* Had administration of another investigational product including vaccines within 60 days or 5 half-lives (whichever is longer), prior to Screening Visit.
* With known history of AIDS or human immunodeficiency virus (HIV) test positive.
* History of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, through medical inquiry.
* History of SARS, SARS-CoV-2 or middle east respiratory syndrome (MERS) infection. Suspected SARS patients should be screened for SARS antibodies.
* Previously participated in a clinical trial involving lipid nanoparticles.
* Are subject to exclusion periods of other clinical trials or simultaneous participation in another clinical trial.
* Have any affiliation with the study site (e.g., are close relative of the investigator or dependent person, such as an employee or student of the study site).
* Have a history of drug abuse or known medical, psychological, or social conditions within the past 5 years. In the opinion of the investigator, could comprise their well-being if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
* Have a history of narcolepsy.
* Have history of alcohol abuse or drug addiction within 1 year prior to Screening Visit.
* Have a history of or suspected immunosuppressive condition, acquired or congenital, as determined by medical history and/or physical examination at Screening Visit.
* Have any abnormality or permanent body art (e.g., tattoo), that in the opinion of the investigator, would obstruct the ability to observe local reactions at the vaccination site.
* Have had any blood loss >400 mL, e.g., due to donation of blood or blood products or injury, within the 28 days prior to Screening Visit or plan to donate blood or plasma during the trial, starting from Screening Visit and continuously until at least 28 days after being given the last immunization.
* Travel or live in any country or region with a high SARS-CoV-2 infection risk (as defined at Screening Visit) within the 14 days prior to Screening Visit.
* They plan to visit any country or region with a high SARS-CoV-2 infection risk (as defined at Screening Visit), from Screening Visit until 14 days after being given the last immunization.
* Symptoms of COVID-19, e.g., respiratory symptoms, fever, cough, shortness of breath and breathing difficulties.
* Have had contact with confirmed COVID-19 patients or persons tested positive for SARS-CoV-2 within the 30 days prior to Screening Visit.
* Are vulnerable persons, e.g., soldiers, subjects in detention, contract research organization (CRO) or Fosun staff or their family members.

For the elderly group (age ≥65 and ≤85)

* Baseline laboratory abnormalities with Grade ≥3 (for hematology abnormalities with Grade ≥2) during screening visits, by physical examination and eligibility screening.
* Have had any acute illness, as determined by the investigator, with or without fever, within 72 hours prior to the prime vaccination. An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the investigator, the residual symptoms will not compromise their well-being if they participate as trial subjects in the trial, or that will not prevent, limit, or confound the protocol-specified assessments.
* Have a known allergy, hypersensitivity, or intolerance to the planned vaccine for trial including any excipients.
* Used to have a history of hypersensitivity or serious reactions to vaccination.
* Received any vaccination within 4 weeks prior to Visit 1.
* Don't agree to not be vaccinated during the trial, starting from Screening Visit and continuously until 28 days after receiving the last immunization, except emergency vaccination (e.g. rabies vaccine, tetanus vaccine).
* Had administration of any immunoglobulins and/or any blood products within the 3 months prior to Screening Visit.
* Had any serious or life-threatening medical condition (e.g., autoimmune disease, cardiovascular disease) within the past 5 years, which in the opinion of the investigator, could compromise their well-being if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
* Have any surgery planned during the trial, starting from Screening Visit and continuously until at least 90 days after the last immunization.
* Had any chronic use (more than 14 continuous days) of any systemic medications that affects immune function, including immunosuppressant or other immune-modifying drugs, within 6 months prior to Screening Visit unless in the opinion of the investigator, the medication would not prevent, limit, or confound the protocol-specified assessments or could compromise safety of subjects.
* Had administration of another investigational product including vaccines within 60 days or 5 half-lives (whichever is longer), prior to Screening Visit.
* With known history of AIDS or HIV test positive.
* History of HBV or HCV infection.
* History of SARS, SARS-CoV-2 or MERS infection. Suspected SARS patients should be screened for SARS antibodies.
* Previously participated in a clinical trial involving lipid nanoparticles.
* Are subject to exclusion periods of other clinical trials or simultaneous participation in another clinical trial.
* Have any affiliation with the study site (e.g., are close relative of the investigator or dependent person, such as an employee or student of the study site).
* Have a history of drug abuse or known medical, psychological, or social conditions within the past 5 years. In the opinion of the investigator, could comprise their well-being if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
* Have a history of narcolepsy.
* Have history of alcohol abuse or drug addiction within 1 year prior to Screening Visit.
* Have a history of or suspected immunosuppressive condition, acquired or congenital, as determined by medical history and/or physical examination at Screening Visit.
* Have any abnormality or permanent body art (e.g., tattoo), that in the opinion of the investigator, would obstruct the ability to observe local reactions at the vaccination site.
* Have had any blood loss >400 mL, e.g., due to donation of blood or blood products or injury, within the 28 days prior to Screening Visit or plan to donate blood or plasma during the trial, starting from Screening Visit and continuously until at least 28 days after being given the last immunization.
* Travel or live in any country or region with a high SARS-CoV-2 infection risk (as defined at Screening Visit) within the 14 days prior to Screening Visit.
* They plan to visit any country or region with a high SARS-CoV-2 infection risk (as defined at Screening Visit), from Screening Visit until 14 days after being given the last immunization.
* Symptoms of COVID-19, e.g., respiratory symptoms, fever, cough, shortness of breath and breathing difficulties.
* Have had contact with confirmed COVID-19 patients or persons tested positive for SARS-CoV-2 nucleic acids or antibodies within the 30 days prior to Screening Visit.
* Are vulnerable persons, e.g., soldiers, subjects in detention, CRO or Fosun staff or their family members.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Taizhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Hui AM, Zhang X, Ge L, Qiu Y, Tang R, Ye H, Wang X, Lin M, Zhu Z, Zheng J, Qiu J, Lagkadinou E, Shpyro S, Ozhelvaci O, Tureci O, Khondker Z, Yin W, Shishkova Y, Jia S, Pan H, Peng F, Ma Z, Wu Z, Guo X, Shi Y, Muik A, Sahin U, Zhu L, Zhu F. Immune Persistence and Safety After SARS-CoV-2 BNT162b1 mRNA Vaccination in Chinese Adults: A Randomized, Placebo-Controlled, Double-Blind Phase 1 Trial. Adv Ther. 2022 Aug;39(8):3789-3798. doi: 10.1007/s12325-022-02206-1. Epub 2022 Jun 30. PMID 35771353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 144 subjects were randomized in this phase I clinical trial, including 72 adult subjects aged 18-55 years old (including boundary value) and 72 elderly subjects aged 65-85 years old (including boundary value). The subjects received either BNT162b1 10 µg (low dose), BNT162b1 30 µg (high dose), or placebo on Day 1 and Day 22, respectively.
Pre-assignment Details: All enrolled participants were allocated to treatment.
Groups:
- Low-dose 10 µg, 18-55 Years of Age; High-dose 30 µg, 18-55 Years of Age; Low-dose 10 µg, 65-85 Years of Age; High-dose 30 µg, 65-85 Years of Age: BNT162b1: Intramuscular injection
Period: Received 2 Doses
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Started | 24 | 24 | 24 | 24 | 24 | 24
Completed | 24 | 24 | 24 | 23 | 23 | 24
Not Completed | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0
Period: Received 2 Doses and Completed Follow-up
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Started | 24 | 24 | 24 | 23 | 23 | 24
Completed | 23 | 24 | 23 | 22 | 22 | 23
Not Completed | 1 | 0 | 1 | 1 | 1 | 1
Not completed — inoculated with other COVID-19 vaccine | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age | Total
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 24 | 0 | 0 | 0 | 72
  >=65 years | 0 | 0 | 0 | 24 | 24 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Totals are presented by age group.
  years
    Group, 18-55 years of age: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0 | 72
    Group, 18-55 years of age | 38 (9.6) | 40 (9.0) | 42 (8.7) |  |  |  | 40 (9.2)
    Group, 65-85 years of age: number analyzed (Participants) | 0 | 0 | 0 | 24 | 24 | 24 | 72
    Group, 65-85 years of age |  |  |  | 71 (5.0) | 69 (3.0) | 71 (4.4) | 70 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 12 | 12 | 12 | 12 | 72
  Male | 12 | 12 | 12 | 12 | 12 | 12 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 24 | 24 | 24 | 24 | 24 | 24 | 144
Region of Enrollment [Number; unit: participants]
  China | 24 | 24 | 24 | 24 | 24 | 24 | 144
Weight [Mean (Standard Deviation); unit: kg] — Population: Totals are presented by age group.
  kg
    Group 18-55 years of age: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0 | 72
    Group 18-55 years of age | 69.5 (12.05) | 62.8 (10.75) | 65.7 (13.26) |  |  |  | 66.0 (12.21)
    Group 65-85 years of age: number analyzed (Participants) | 0 | 0 | 0 | 24 | 24 | 24 | 72
    Group 65-85 years of age |  |  |  | 61.8 (9.83) | 63.8 (8.81) | 59.0 (8.36) | 61.5 (9.11)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Totals are presented by age group.
  kg/m^2
    Group 18-55 years of age: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0 | 72
    Group 18-55 years of age | 24.7 (3.18) | 23.0 (2.71) | 24.3 (3.43) |  |  |  | 24.0 (3.16)
    Group 65-85 years of age: number analyzed (Participants) | 0 | 0 | 0 | 24 | 24 | 24 | 72
    Group 65-85 years of age |  |  |  | 23.9 (2.95) | 24.8 (2.85) | 23.5 (2.45) | 24.1 (2.77)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) (e.g., Injection Site Pain, Redness, Induration, Swelling) Recorded up to 14 Days After Each Dose of BNT162b1 or Placebo.
Description: Solicited local AEs were collected within 7 days/14 days after each vaccination. For the grading of AEs, a 7-day period AE assessment after each dose as graded by United States (US) Food and Drug Administration (FDA) criteria along with the 14-day period AE assessment as graded by National Medical Products Administration (NMPA) criteria are used to evaluate solicited AEs. For other AEs, only the NMPA criteria is used. The "solicited" AEs were pre-defined and listed in the subjects' diaries. All the solicited local AEs occurred within 7 days after vaccination were related to investigational vaccine (or placebo).
Time Frame: Up to 14 days following each dose administration
Population: Safety Analysis Set including all randomized participants who receive at least one dose of the investigational vaccine/placebo and at least one safety evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Within 7 days after dose 1: Number of participants with solicited local AEs | 19 | 24 | 1 | 13 | 19 | 0
  Within 7 days after dose 2: Number of participants with solicited local AEs | 17 | 20 | 1 | 15 | 15 | 0
  Within 7 days after dose 1: Number of participants with solicited local AEs grade 3 (FDA criteria) | 0 | 0 | 0 | 0 | 0 | 0
  Within 7 days after dose 2: Number of participants with solicited local AEs grade 3 (FDA criteria) | 0 | 0 | 0 | 0 | 0 | 0
  Within 14 days after dose 1: Number of participants with solicited local AEs grade 3 (NMPA criteria) | 0 | 0 | 0 | 0 | 0 | 0
  Within 14 days after dose 2: Number of participants with solicited local AEs grade 3 (NMPA criteria) | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Solicited Systemic AEs (e.g., e.g., Nausea, Vomiting, Diarrhea, Headache, Fatigue, Myalgia, Arthralgia, Chills, Loss of Appetite, Malaise, and Fever) Recorded up to 14 Days After Each Dose of BNT162b1 or Placebo.
Description: Solicited systemic AEs were collected within 7 days/14 days after each vaccination. For the grading of AEs, a 7-day period AE assessment after each dose as graded by US FDA criteria along with the 14-day period AE assessment as graded by NMPA criteria are used to evaluate solicited AEs. For other AEs, only the NMPA criteria is used. The "solicited" AEs were pre-defined and listed in the subjects' diaries. Except for 1 event (myalgia) occurred in 10 µg group and 1 event (diarrhea) occurred in placebo group, all the solicited systemic AEs occurred within 7 days after vaccination were related to investigational vaccine (or placebo). All the solicited systemic AEs occurred within 14 days after vaccination were related to investigational vaccine (or placebo), except for 1 event (myalgia) occurred in placebo group and 2 events (both diarrhea; 1 event occurred in 30 µg group, 1 event occurred in placebo group).
Time Frame: Up to 14 days following each dose administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Within 7 d (days) after dose 1: Number of participants with solicited systemic AEs | 9 | 16 | 3 | 3 | 15 | 2
  Within 7 d after dose 2: Number of participants with solicited systemic AEs | 15 | 21 | 3 | 7 | 17 | 1
  Within 14 d after dose 1: Number of participants with solicited systemic AEs | 10 | 16 | 3 | 3 | 15 | 2
  Within 14 d after dose 2: Number of participants with solicited systemic AEs | 15 | 21 | 3 | 7 | 17 | 2
  Within 7 d after dose 1: Number of participants with related solicited systemic AEs grade 3 (FDA) | 0 | 1 | 0 | 0 | 2 | 0
  Within 7 d after dose 2: Number of participants with related solicited systemic AEs grade 3 (FDA) | 1 | 3 | 0 | 0 | 0 | 0
  Within 14 d after dose 1: Number of participants with related solicited systemic AEs grade 3 (NMPA) | 0 | 5 | 0 | 0 | 2 | 0
  Within 14 d after dose 2: Number of participants with related solicited systemic AEs grade 3 (NMPA) | 3 | 6 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Unsolicited Vaccine Related AEs During the 21-day Period After Dose 1 of BNT162b1 or Placebo.
Description: AEs occurred during the 21-day period after dose 1 were also referred as "unsolicited" AEs. The unsolicited AEs were not pre-defined in the subjects' diaries.
Time Frame: 21-day period after dose 1 vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
participants | 7 | 7 | 1 | 2 | 5 | 2

4. Primary Outcome: Number of Participants With Unsolicited Vaccine Related AEs During the 28-day Period After Dose 2 of BNT162b1 or Placebo.
Description: AEs occurred during the 28-day period after dose 2 were also referred as "unsolicited" AEs. The unsolicited AEs were not pre-defined in the subjects' diaries.
Time Frame: 28-day period after dose 2 vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
participants | 5 | 8 | 0 | 2 | 7 | 0

5. Secondary Outcome: The Number of Participants Experiencing Treatment Emergent Serious Adverse Events (TESAEs)
Time Frame: From Dose 1 up to Month 12
Population: Safety Analysis Set including all randomized subjects who receive at least one dose of the investigational vaccine/placebo and at least one safety evaluation.
Measure: Number; unit: participants
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
participants | 0 | 1 | 1 | 1 | 0 | 0

6. Secondary Outcome: The Number of Participants Experiencing Related TEAEs
Description: "Related" implies the relationship between AE and vaccine is one of "Possibly related", "Probably related" and "Definitely related".
Time Frame: From Dose 1 up to Month 12
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
participants
  Number of Participants with related TEAEs after dose 1 | 22 | 24 | 4 | 16 | 21 | 4
  Number of Participants with related TEAEs after dose 2 | 20 | 22 | 4 | 18 | 21 | 0

7. Secondary Outcome: The Number of Participants Experiencing Clinically Significant (CS) Abnormal Markers of Hematology, Blood Chemistry and Urine Analysis
Description: Results for CS results are displayed by abnormal parameter. Abnormal test results assessed not clinical significant are not presented. Participants with more than one 'CS' parameter are counted for each parameter separately and therefore included multiple times.
Time Frame: Hour 24 and Day 7 after dose 1 and Day 7 after dose 2
Population: The safety analysis set included all randomized subjects who receive at least one dose of the investigational vaccine/placebo and have at least one safety evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Participants
  CS abnormal blood chemistry parameter - increased total bilirubin - 24 hours after dose 1 | 0 | 1 | 0 | 0 | 0 | 0
  CS abnormal blood chemistry parameter - increased total bilirubin - Day 7 after dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal blood chemistry parameter - increased total bilirubin - Day 7 after dose 2: number analyzed (Participants) | 24 | 24 | 24 | 23 | 23 | 24
  CS abnormal blood chemistry parameter - increased total bilirubin - Day 7 after dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal urine routine test results - elevated leucocyte (microscopic) - 24 hours after dose 1 | 1 | 0 | 1 | 0 | 0 | 1
  CS abnormal urine routine test results - elevated leucocyte (microscopic) - Day 7 after dose 1 | 0 | 0 | 0 | 1 | 0 | 0
  CS abnormal urine routine test results - elevated leucocyte (microscopic) - Day 7 after dose 2: number analyzed (Participants) | 24 | 24 | 24 | 23 | 22 | 24
  CS abnormal urine routine test results - elevated leucocyte (microscopic) - Day 7 after dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal urine routine test results - bacteria (microscopic) - 24 hours after dose 1 | 1 | 0 | 1 | 0 | 0 | 1
  CS abnormal urine routine test results - bacteria (microscopic) - Day 7 after dose 1 | 0 | 0 | 0 | 1 | 0 | 1
  CS abnormal urine routine test results - bacteria (microscopic) - Day 7 after dose 2: number analyzed (Participants) | 24 | 24 | 24 | 23 | 22 | 24
  CS abnormal urine routine test results - bacteria (microscopic) - Day 7 after dose 2 | 0 | 0 | 0 | 1 | 0 | 0
  CS abnormal urine routine test results - red blood cells (microscopic) - 24 hours after dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal urine routine test results - red blood cells (microscopic) - Day 7 after dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal urine routine test results - red blood cells (microscopic) - Day 7 after dose 2: number analyzed (Participants) | 24 | 24 | 24 | 23 | 22 | 24
  CS abnormal urine routine test results - red blood cells (microscopic) - Day 7 after dose 2 | 0 | 0 | 0 | 1 | 0 | 0
  CS abnormal urine routine test results - glucose - 24 hours after dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal urine routine test results - glucose - Day 7 after dose 1 | 0 | 0 | 0 | 0 | 1 | 0
  CS abnormal urine routine test results - glucose - Day 7 after dose 2: number analyzed (Participants) | 24 | 24 | 24 | 23 | 22 | 24
  CS abnormal urine routine test results - glucose - Day 7 after dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal urine routine test results - ketone - 24 hours after dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal urine routine test results - ketone - Day 7 after dose 1 | 0 | 0 | 0 | 0 | 1 | 0
  CS abnormal urine routine test results - ketone - Day 7 after dose 2: number analyzed (Participants) | 24 | 24 | 24 | 23 | 22 | 24
  CS abnormal urine routine test results - ketone - Day 7 after dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal urine routine test results - blood - 24 hours after dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal urine routine test results - blood - Day 7 after dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal urine routine test results - blood - Day 7 after dose 2: number analyzed (Participants) | 24 | 24 | 24 | 23 | 22 | 24
  CS abnormal urine routine test results - blood - Day 7 after dose 2 | 0 | 0 | 0 | 1 | 0 | 0
  CS abnormal hematology parameter - hemoglobin - 24 hours after dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal hematology parameter - hemoglobin - Day 7 after dose 1 | 1 | 0 | 0 | 0 | 0 | 0
  CS abnormal hematology parameter - hemoglobin - Day 7 after dose 2: number analyzed (Participants) | 24 | 24 | 24 | 23 | 23 | 24
  CS abnormal hematology parameter - hemoglobin - Day 7 after dose 2 | 1 | 1 | 0 | 0 | 0 | 0
  CS abnormal hematology parameter - hematocrit - 24 hours after dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal hematology parameter - hematocrit - Day 7 after dose 1 | 1 | 0 | 0 | 0 | 0 | 0
  CS abnormal hematology parameter - hematocrit - Day 7 after dose 2: number analyzed (Participants) | 24 | 24 | 24 | 23 | 23 | 24
  CS abnormal hematology parameter - hematocrit - Day 7 after dose 2 | 1 | 1 | 0 | 0 | 0 | 0
  CS abnormal hematology parameter - lymphocyte - 24 hours after dose 1 | 3 | 5 | 0 | 0 | 0 | 0
  CS abnormal hematology parameter - lymphocyte - Day 7 after dose 1 | 0 | 0 | 0 | 0 | 0 | 1
  CS abnormal hematology parameter - lymphocyte - Day 7 after dose 2: number analyzed (Participants) | 24 | 24 | 24 | 23 | 22 | 24
  CS abnormal hematology parameter - lymphocyte - Day 7 after dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  CS abnormal hematology parameter - platelet count - 24 hours after dose 1 | 0 | 2 | 0 | 1 | 2 | 0
  CS abnormal hematology parameter - platelet count - Day 7 after dose 1 | 0 | 0 | 1 | 1 | 0 | 0
  CS abnormal hematology parameter - platelet count - Day 7 after dose 2: number analyzed (Participants) | 24 | 24 | 24 | 23 | 23 | 24
  CS abnormal hematology parameter - platelet count - Day 7 after dose 2 | 0 | 0 | 2 | 1 | 0 | 0

8. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-S1 IgG Antibody
Description: At Day 7, Day 21 after dose 1, at Day 7, Day 21 after dose 2, and at Month 3, 6 and 12 after dose 1.
Time Frame: Up to 12 months following first dose
Population: Per Protocol Set (PPS) - all subjects in the Total Vaccinated Cohort (TVC) who had no major protocol violations and completed dose 2. The TVC included all randomized subjects who had received at least one dose of the investigational vaccine/placebo and could provide with effective baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 23 | 24
titer
  7 days after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  7 days after dose 1 | 53.320 [46.680 to 60.905] | 59.220 [41.728 to 84.046] | 52.841 [47.132 to 59.242] |  |  |
  21 days after dose 1 | 4193.710 [2664.050 to 6601.681] | 4531.416 [3029.130 to 6778.757] | 52.594 [47.369 to 58.395] | 859.646 [467.549 to 1580.564] | 2872.861 [1685.729 to 4896.002] | 62.239 [47.583 to 81.410]
  7 days after dose 2 | 26548.853 [18381.541 to 38345.078] | 41530.498 [33984.171 to 50752.518] | 52.578 [47.384 to 58.341] | 5271.560 [2484.575 to 11184.748] | 23447.197 [15268.301 to 36007.348] | 62.658 [47.633 to 82.423]
  21 days after dose 2 | 46810.469 [41673.251 to 52580.970] | 49773.381 [46947.113 to 52769.794] | 50.000 [50.000 to 50.000] | 40942.862 [33177.420 to 50525.869] | 44159.581 [37139.275 to 52506.910] | 61.008 [45.725 to 81.399]
  Month 3 after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  Month 3 after dose 1 | 27143.015 [21023.440 to 35043.897] | 31584.450 [26378.938 to 37817.196] | 50.000 [50.000 to 50.000] |  |  |
  Month 6 after dose 1: number analyzed (Participants) | 24 | 24 | 22 | 23 | 23 | 23
  Month 6 after dose 1 | 4169.448 [2978.898 to 5835.815] | 5693.082 [4412.125 to 7345.934] | 55.088 [47.853 to 63.417] | 2223.699 [1565.907 to 3157.811] | 4970.376 [3625.506 to 6814.121] | 60.931 [45.837 to 80.995]
  Month 12 after dose 1: number analyzed (Participants) | 23 | 24 | 23 | 22 | 22 | 23
  Month 12 after dose 1 | 2002.152 [1389.905 to 2884.090] | 2792.605 [2118.269 to 3681.610] | 50.000 [50.000 to 50.000] | 1104.860 [698.932 to 1746.542] | 2847.010 [1887.353 to 4294.621] | 53.105 [46.867 to 60.174]

9. Secondary Outcome: GMT of Anti-receptor Binding Domain (RBD) Immunoglobulin G (IgG) Antibody
Description: At Day 7, Day 21 after dose 1, at Day 7, Day 21 after dose 2, and at Month 3, 6 and 12 after dose 1.
Time Frame: Up to 12 months following first dose
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 23 | 24
titer
  7 days after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  7 days after dose 1 | 50.000 [50.000 to 50.000] | 52.903 [47.074 to 59.453] | 56.644 [48.999 to 65.482] |  |  |
  21 days after dose 1 | 13095.167 [8395.009 to 20426.827] | 13046.378 [8950.882 to 19015.777] | 56.699 [49.052 to 65.537] | 3040.808 [1569.768 to 5890.369] | 10370.854 [5955.358 to 18060.142] | 74.476 [55.679 to 99.618]
  7 days after dose 2 | 38314.550 [30173.509 to 48652.107] | 47324.691 [43213.653 to 51826.824] | 57.377 [49.028 to 67.146] | 10748.566 [5512.317 to 20958.821] | 38256.083 [30078.753 to 48656.534] | 75.817 [55.962 to 102.715]
  21 days after dose 2 | 49710.291 [46764.743 to 52841.369] | 51200.000 [51200.000 to 51200.000] | 60.605 [48.454 to 75.804] | 46980.825 [42021.855 to 52525.000] | 50977.162 [50528.938 to 51429.363] | 65.756 [53.237 to 81.218]
  Month 3 after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  Month 3 after dose 1 | 40236.195 [32999.573 to 49059.768] | 43050.715 [38767.819 to 47806.766] | 60.439 [49.911 to 73.188] |  |  |
  Month 6 after dose 1: number analyzed (Participants) | 24 | 24 | 22 | 23 | 23 | 23
  Month 6 after dose 1 | 8249.604 [6186.091 to 11001.449] | 9608.488 [7410.049 to 12459.167] | 61.768 [50.272 to 75.894] | 4114.353 [2716.614 to 6231.250] | 7187.827 [5138.636 to 10054.194] | 54.780 [48.060 to 62.439]
  Month 12 after dose 1: number analyzed (Participants) | 23 | 24 | 23 | 22 | 22 | 23
  Month 12 after dose 1 | 2324.072 [1677.862 to 3219.163] | 2804.882 [2191.409 to 3590.094] | 56.083 [47.501 to 66.216] | 1536.143 [921.738 to 2560.094] | 2768.366 [1880.754 to 4074.881] | 63.175 [50.876 to 78.447]

10. Secondary Outcome: GMT of SARS-CoV-2 Neutralizing Antibody (Including True Virus-based SARS-CoV-2 Neutralizing Test)
Description: At Day 7, Day 21 after first dose, at Day 7, Day 21 after second dose, and at Month 3, 6, and 12 after first dose.
Time Frame: Up to 12 months following first dose
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 23 | 24
titer
  7 days after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  7 days after dose 1 | 5.000 [5.000 to 5.000] | 5.000 [5.000 to 5.000] | 5.000 [5.000 to 5.000] |  |  |
  21 days after dose 1 | 18.877 [10.586 to 33.664] | 14.557 [9.712 to 21.817] | 5.000 [5.000 to 5.000] | 6.965 [5.037 to 9.633] | 10.946 [7.213 to 16.612] | 5.000 [5.000 to 5.000]
  7 days after dose 2 | 56.569 [31.503 to 101.579] | 119.865 [81.547 to 176.187] | 5.000 [5.000 to 5.000] | 14.357 [8.689 to 23.721] | 49.394 [26.334 to 92.647] | 5.000 [5.000 to 5.000]
  21 days after dose 2 | 232.905 [151.299 to 358.525] | 253.984 [184.601 to 349.445] | 5.000 [5.000 to 5.000] | 80.000 [49.173 to 130.153] | 160.000 [96.736 to 264.637] | 5.000 [5.000 to 5.000]
  Month 3 after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  Month 3 after dose 1 | 54.958 [38.115 to 79.245] | 87.241 [64.445 to 118.099] | 5.000 [5.000 to 5.000] |  |  |
  Month 6 after dose 1: number analyzed (Participants) | 24 | 24 | 22 | 23 | 23 | 23
  Month 6 after dose 1 | 16.339 [11.274 to 23.679] | 27.479 [20.383 to 37.046] | 5.000 [5.000 to 5.000] | 10.000 [7.219 to 13.852] | 20.612 [13.303 to 31.937] | 5.000 [5.000 to 5.000]
  Month 12 after dose 1: number analyzed (Participants) | 23 | 24 | 23 | 22 | 22 | 23
  Month 12 after dose 1 | 7.858 [6.027 to 10.244] | 11.892 [8.903 to 15.885] | 5.000 [5.000 to 5.000] | 6.040 [4.976 to 7.333] | 12.081 [8.154 to 17.899] | 5.000 [5.000 to 5.000]

11. Secondary Outcome: Fold Increase in Antibody Anti-S1 IgG Antibody Titers, as Compared to Baseline
Description: At Day 7, Day 21 after dose 1, at Day 7, Day 21 after dose 2, and at Month 3, 6, and 12 after dose 1.
Time Frame: Up to 12 months following the first dose
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 23 | 24
fold rise
  7 days after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  7 days after dose 1 | 0.960 [0.899 to 1.025] | 0.998 [0.993 to 1.002] | 0.992 [0.976 to 1.008] |  |  |
  21 days after dose 1 | 75.535 [45.607 to 125.103] | 76.351 [48.641 to 119.845] | 0.988 [0.962 to 1.013] | 16.501 [8.998 to 30.260] | 52.377 [30.969 to 88.586] | 0.997 [0.991 to 1.002]
  7 days after dose 2 | 478.186 [316.204 to 723.147] | 699.755 [473.456 to 1034.219] | 0.987 [0.961 to 1.014] | 101.189 [47.897 to 213.776] | 427.484 [281.104 to 650.090] | 1.003 [0.998 to 1.008]
  21 days after dose 2 | 843.129 [696.113 to 1021.194] | 838.640 [586.916 to 1198.328] | 0.939 [0.824 to 1.070] | 785.911 [631.437 to 978.175] | 805.108 [655.534 to 988.810] | 0.977 [0.896 to 1.065]
  Month 3 after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  Month 3 after dose 1 | 488.888 [359.289 to 665.234] | 532.172 [371.322 to 762.699] | 0.939 [0.824 to 1.070] |  |  |
  Month 6 after dose 1: number analyzed (Participants) | 24 | 24 | 22 | 23 | 23 | 23
  Month 6 after dose 1 | 75.098 [50.105 to 112.558] | 95.924 [66.863 to 137.614] | 1.028 [0.939 to 1.126] | 42.685 [29.500 to 61.762] | 90.619 [64.457 to 127.399] | 0.966 [0.886 to 1.054]
  Month 12 after dose 1: number analyzed (Participants) | 23 | 24 | 23 | 22 | 22 | 23
  Month 12 after dose 1 | 35.898 [23.326 to 55.246] | 47.053 [33.587 to 65.918] | 0.936 [0.817 to 1.073] | 21.169 [13.164 to 34.039] | 51.688 [34.959 to 76.423] | 0.842 [0.664 to 1.069]

12. Secondary Outcome: Fold Increase in Antibody Anti-RBD IgG Antibody Titers, as Compared to Baseline
Description: At Day 7, Day 21 after dose 1, at Day 7, Day 21 after dose 2, and at Month 3, 6, and 12 after dose 1.
Time Frame: Up to 12 months following first dose
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 23 | 24
fold rise
  7 days after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  7 days after dose 1 | 1.000 [1.000 to 1.000] | 1.001 [0.998 to 1.005] | 0.985 [0.968 to 1.003] |  |  |
  21 days after dose 1 | 261.903 [167.900 to 408.537] | 246.976 [172.957 to 352.672] | 0.986 [0.964 to 1.009] | 51.597 [28.409 to 93.710] | 150.858 [74.500 to 305.479] | 1.001 [0.985 to 1.018]
  7 days after dose 2 | 766.291 [603.470 to 973.042] | 895.886 [778.927 to 1030.407] | 0.998 [0.973 to 1.023] | 182.382 [96.770 to 343.735] | 556.487 [351.897 to 880.024] | 1.020 [0.981 to 1.059]
  21 days after dose 2 | 994.206 [935.295 to 1056.827] | 969.249 [865.101 to 1085.934] | 1.054 [0.990 to 1.122] | 797.173 [645.312 to 984.773] | 741.532 [498.207 to 1103.699] | 0.884 [0.753 to 1.038]
  Month 3 after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  Month 3 after dose 1 | 804.724 [659.991 to 981.195] | 814.977 [706.611 to 939.963] | 1.051 [0.970 to 1.140] |  |  |
  Month 6 after dose 1: number analyzed (Participants) | 24 | 24 | 22 | 23 | 23 | 23
  Month 6 after dose 1 | 164.992 [123.722 to 220.029] | 181.895 [145.883 to 226.796] | 1.061 [0.889 to 1.267] | 69.813 [47.788 to 101.988] | 104.557 [65.750 to 166.268] | 0.764 [0.615 to 0.950]
  Month 12 after dose 1: number analyzed (Participants) | 23 | 24 | 23 | 22 | 22 | 23
  Month 12 after dose 1 | 46.481 [33.557 to 64.383] | 53.098 [42.807 to 65.863] | 0.970 [0.893 to 1.053] | 25.871 [16.436 to 40.724] | 41.548 [25.869 to 66.729] | 0.835 [0.690 to 1.010]

13. Secondary Outcome: Fold Increase in SARS-CoV-2 Neutralizing Antibody Titers (Virus Neutralizing Test), as Compared to Baseline.
Description: At Day 7, Day 21 after dose 1, at Day 7, Day 21 after dose 2, and at Month 3, 6, and 12 after dose 1.
Time Frame: Up to 12 months following first dose
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 23 | 24
fold rise
  7 days after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  7 days after dose 1 | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000] | 1.000 [1.000 to 1.000] |  |  |
  21 days after dose 1 | 3.775 [2.117 to 6.733] | 2.911 [1.942 to 4.363] | 1.000 [1.000 to 1.000] | 1.393 [1.007 to 1.927] | 2.189 [1.443 to 3.322] | 1.000 [1.000 to 1.000]
  7 days after dose 2 | 11.314 [6.301 to 20.316] | 23.973 [16.309 to 35.237] | 1.000 [1.000 to 1.000] | 2.871 [1.738 to 4.744] | 9.879 [5.267 to 18.529] | 1.000 [1.000 to 1.000]
  21 days after dose 2 | 46.581 [30.260 to 71.705] | 50.797 [36.920 to 69.889] | 1.000 [1.000 to 1.000] | 16.000 [9.835 to 26.031] | 32.000 [19.347 to 52.927] | 1.000 [1.000 to 1.000]
  Month 3 after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  Month 3 after dose 1 | 10.992 [7.623 to 15.849] | 17.448 [12.889 to 23.620] | 1.000 [1.000 to 1.000] |  |  |
  Month 6 after dose 1: number analyzed (Participants) | 24 | 24 | 22 | 23 | 23 | 23
  Month 6 after dose 1 | 3.268 [2.255 to 4.736] | 5.496 [4.077 to 7.409] | 1.000 [1.000 to 1.000] | 2.000 [1.444 to 2.770] | 4.122 [2.661 to 6.387] | 1.000 [1.000 to 1.000]
  Month 12 after dose 1: number analyzed (Participants) | 23 | 24 | 23 | 22 | 22 | 23
  Month 12 after dose 1 | 1.572 [1.205 to 2.049] | 2.378 [1.781 to 3.177] | 1.000 [1.000 to 1.000] | 1.208 [0.995 to 1.467] | 2.416 [1.631 to 3.580] | 1.000 [1.000 to 1.000]

14. Secondary Outcome: Seroconversion Rates (SCR) Defined as a Minimum of 4-fold Increase of Antibody Titers, as Compared to Baseline
Description: At Day 7, Day 21 after dose 1, and at Day 7, Day 21 after dose 2.
Time Frame: Up to 21 days after dose 2
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
Number analyzed (Participants) | 24 | 24 | 24 | 23 | 23 | 24
Participants
  SCR of SARS-CoV-2 neutralizing antibody - 7 days after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  SCR of SARS-CoV-2 neutralizing antibody - 7 days after dose 1 | 0 | 0 | 0 |  |  |
  SCR of SARS-CoV-2 neutralizing antibody - 21 days after dose 1 | 12 | 11 | 0 | 3 | 8 | 0
  SCR of SARS-CoV-2 neutralizing antibody - 7 days after dose 2 | 18 | 23 | 0 | 11 | 18 | 0
  SCR of SARS-CoV-2 neutralizing antibody - 21 days after dose 2 | 24 | 24 | 0 | 21 | 22 | 0
  SCR of anti-S1 IgG antibody - 7 days after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  SCR of anti-S1 IgG antibody - 7 days after dose 1 | 0 | 0 | 0 |  |  |
  SCR of anti-S1 IgG antibody - 21 days after dose 1 | 24 | 24 | 0 | 21 | 22 | 0
  SCR of anti-S1 IgG antibody - 7 days after dose 2 | 24 | 24 | 0 | 22 | 23 | 0
  SCR of anti-S1 IgG antibody - 21 days after dose 2 | 24 | 24 | 0 | 23 | 23 | 0
  SCR of anti-RBD IgG antibody - 7 days after dose 1: number analyzed (Participants) | 24 | 24 | 24 | 0 | 0 | 0
  SCR of anti-RBD IgG antibody - 7 days after dose 1 | 0 | 0 | 0 |  |  |
  SCR of anti-RBD IgG antibody - 21 days after dose 1 | 24 | 24 | 0 | 22 | 22 | 0
  SCR of anti-RBD IgG antibody - 7 days after dose 2 | 24 | 24 | 0 | 23 | 23 | 0
  SCR of anti-RBD IgG antibody - 21 days after dose 2 | 24 | 24 | 0 | 23 | 23 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 (Dose 1) up to last visit (approximately 12 months after first dose)
Description: Treatment-emergent AEs (TEAEs) are presented, including solicited and unsolicited AEs.
  An TEAE is defined as any AE with an onset date on or after the first dose (if the AE was absent before the first dose) or worsened after the first dose (if the AE was present before the first dose). AEs with an onset date more than 28 days after the last dose will be considered as treatment emergent only if assessed as related to the vaccine (BNT162b1 or placebo) by the investigator.
Arm/Group | Low-dose 10 µg, 18-55 Years of Age | High-dose 30 µg, 18-55 Years of Age | Placebo, 18-55 Years of Age | Low-dose 10 µg, 65-85 Years of Age | High-dose 30 µg, 65-85 Years of Age | Placebo, 65-85 Years of Age
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/24 | 1/24 | 1/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 22/24 | 24/24 | 7/24 | 22/24 | 24/24 | 9/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose 10 µg, 18-55 Years of Age (N=24) | High-dose 30 µg, 18-55 Years of Age (N=24) | Placebo, 18-55 Years of Age (N=24) | Low-dose 10 µg, 65-85 Years of Age (N=24) | High-dose 30 µg, 65-85 Years of Age (N=24) | Placebo, 65-85 Years of Age (N=24)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose 10 µg, 18-55 Years of Age (N=24) | High-dose 30 µg, 18-55 Years of Age (N=24) | Placebo, 18-55 Years of Age (N=24) | Low-dose 10 µg, 65-85 Years of Age (N=24) | High-dose 30 µg, 65-85 Years of Age (N=24) | Placebo, 65-85 Years of Age (N=24)
Vaccination site pain (General disorders) | 21 (36) | 23 (42) | 2 (2) | 16 (25) | 21 (34) | 0 (0)
Pyrexia (General disorders) | 14 (14) | 21 (33) | 1 (1) | 7 (8) | 19 (31) | 1 (1)
Fatigue (General disorders) | 13 (16) | 16 (23) | 0 (0) | 3 (3) | 8 (10) | 0 (0)
Malaise (General disorders) | 8 (8) | 9 (12) | 0 (0) | 2 (2) | 4 (5) | 1 (1)
Vaccination site erythema (General disorders) | 6 (7) | 8 (11) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
Vaccination site swelling (General disorders) | 5 (5) | 7 (9) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Chills (General disorders) | 4 (4) | 7 (9) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Temperature intolerance (General disorders) | 2 (2) | 6 (7) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Vaccination site discomfort (General disorders) | 3 (4) | 4 (4) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
Vaccination site pruritus (General disorders) | 2 (3) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site induration (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 11 (12) | 19 (25) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 6 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (14) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 10 (14) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs respectively trial sites shall not publish or refer to in writing or orally, in whole or in part, any data, information or materials generated from the study and the services, without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT04523571/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT04523571/SAP_001.pdf